CLINICAL TRIAL: NCT06670053
Title: Effect of Testosterone on Brain Imaging and Headache in Transmasculine Adolescents
Brief Title: Puberty, Testosterone, and Brain Development
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 23-1113
Record Dates: First submitted 2024-10-23; First posted 2024-11-01 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Gender Identity; Gender Dysphoria in Adolescents and Adults; Headache; Transgender
Keywords: resting-state functional connectivity; pain task; fMRI; MRI; migraine; gender affirming hormone therapy; testosterone
MeSH Terms: conditions — Headache; Migraine Disorders | interventions — Testosterone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- On blocker: Transmasculine youth who will begin taking testosterone clinically in < 6 months with or without headache and who have been on pubertal blocker, a gonadotropin hormone releasing (GnRH) agonist for at least 3 months.
  Interventions: Drug: Testosterone
- No blocker: Transmasculine youth who will begin taking testosterone clinically in < 6 months with or without headache and who have no history of pubertal blocker.
  Interventions: Drug: Testosterone

INTERVENTIONS:
Drug: Testosterone — Clinical testosterone therapy
  No research interventions will be used as a part of the study since the research is observational. Testosterone treatment will be prescribed and followed by participant's clinical physician.

SUMMARY:
Transmasculine youth (female sex assigned at birth, male gender identity) who begin clinical gender affirming hormone therapy (GAHT) with testosterone (T) may experience changes in headache. Researchers think this because studies published on effects of giving testosterone to cisgender females (female sex, female gender identity) and transmasculine adults seem to show an effect on pain.

This research will help us learn more about changes in headache and in brain structure and function in transmasculine youth during the first two years of T. Youth who will be starting T within 6 months, either on puberty blocker or not, as part of their regular medical care can participate and will be asked to attend 4 visits:

* before starting T
* after 6 months on T
* after 1 year on T
* after 2 years on T

At the visits, they will be asked to:

* answer questions and surveys about their health
* have a brain MRI done
* give a small sample of blood

and at their first visit, complete a physical exam. Some participants can also do a brief test of pain sensitivity. All participants will be asked to complete a headache diary for the first 6 months, for 1 month after the 1 year visit, and for 1 month after the 2 year visit.

DETAILED DESCRIPTION:
This will be conducted at Childrens Hospital Colorado (CHCO) Clinical & Translational Research Centers (CTRC) facilities. Physical examination will include vital signs, anthropometric measurements, and breast/pubic hair staging, as applicable, by a medical provider.

Visits will be in the morning to capture peak hormone levels.

The following questionnaires will be administered: PROMIS Pediatric Anxiety Short Form, PROMIS Pediatric Depressive Symptoms Short Form, and PedMIDAS form (headache disability measure).

The daily headache diary is tailored to be brief on days when no headache occurs, and to capture more detail including medications taken and headache and aura characteristics on days a headache does occur.

The medical chart will be reviewed for relevant health information and medications.

MR-based imaging will be conducted at the Brain Imaging Center at the University of Colorado Anschutz Medical Campus.

ELIGIBILITY:
Inclusion Criteria:

1. transmasculine and gender diverse
2. assigned female at birth
3. age 12-20 years at the time of enrollment
4. plan to start testosterone clinically in < 6 months
5. if taking gonadotropin releasing hormone agonist (GnRHa, puberty blocker), was started on this type of drug 3+ months prior to enrollment

Exclusion Criteria:

1. cognitive or psychiatric impairment resulting in inability to tolerate or perform the study procedures
2. known history of stroke, multiple sclerosis, or other serious neurologic condition
3. prior diagnosis of Turner Syndrome (monosomy X) or other difference of sexual development
4. prior diagnosis of polycystic ovarian syndrome (PCOS)
5. uncontrolled or untreated hypothyroidism
6. MRI-specific exclusion criteria: (Weight > 500 lbs, severe claustrophobia, certain type of metal in body)

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Transmasculine, gender diverse
Study Population: transmasculine and gender diverse youth
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-31 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in headache burden | Over the two years of the study
  Change in number of headache days per month
Amygdala volume | At the end of the two years of study
  As measured by volumetric MRI

SECONDARY OUTCOMES:
Headache diagnosis | At baseline visit before start of T
  Application of ICHD-3 criteria to headaches, if any

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Hranilovich, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No